CLINICAL TRIAL: NCT06792305
Title: SEQUENCE OF FIXATION IN VERTICALLY UNSTABLE TILE C1.2 AND C1.3 PELVIC RING INJURIES: A PROSPECTIVE COMPARATIVE STUDY
Brief Title: The Sequence of Fixation in Tile C1.2 and C1.3 Vertical Shear Pelvic Ring Injuries.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Karim Atef Salem, Dr, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU R230/2024; No funds recieved (Other: Ainshams University)
Record Dates: First submitted 2024-11-23; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Ring Fractures; Pelvic Ring Injury
Keywords: pelvic ring injuries; vertical shear pelvic fracture; tile classification

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A will be fixed anteriorly first (Active Comparator): Group A will consist of 15 patients and will be fixed anteriorly first.
  Interventions: Procedure: Starting by anterior ring fixation in vertical shear pelvic ring injuries
- Group B will be fixed posteriorly first (Active Comparator): Group B: 15 cases, and will be fixed posteriorly first.
  Interventions: Procedure: Starting by posterior ring fixation in vertical shear pelvic ring injuries

INTERVENTIONS:
Procedure: Starting by anterior ring fixation in vertical shear pelvic ring injuries — The procedure will involve addressing the pelvic ring anteriorly with open reduction and internal fixation (ORIF) of the pubic rami and symphysis pubis by using a single 3.5 mm recon plate. The goal isto achieve anatomical reduction and stable fixation to restore the integrity of the pelvic ring. Fixation of the posterior ring will be achieved using a single sacroiliac screw in S1. The goal of posterior fixation is to achieve stability and alignment of the posterior pelvic structures.
  Arms: Group A will be fixed anteriorly first
Procedure: Starting by posterior ring fixation in vertical shear pelvic ring injuries — the procedure will involve fixation of the posterior ring which will be achieved by using a single sacroiliac screw in S1. Then open reduction and internal fixation (ORIF) of the pubic rami and symphysis pubis by using a single 3.5 mm recon plate.
  Arms: Group B will be fixed posteriorly first

SUMMARY:
The goal of this study is to compare the sequence of fixation in Vertically Unstable Tile C1.2 and C1.3 pelvic ring injuries, as regards clinical, radiological outcomes and implant failure rates. Our hypothesis is that starting with anterior ring fixation will achieve superior results as regards easier reduction, less operation time, and finally better radiological and functional outcomes when compared with starting with posterior ring fixation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years - 60 years.
2. Tile C1.2 and C1.3 pelvic ring injuries.
3. Pure anterior ring ligamentous injuries.

Exclusion Criteria:

1. Bony fracture of the pubic rami.
2. Tile C2 and C3 pelvic ring injuries.
3. Associated acetabular fracture that requires intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Radiological outcome scores | 12 months
  Patients will be followed up at two weeks, six weeks, three months, six months and one year postoperatively. Matta & Tornetta radiological principles will be used to assess the radiological and clinical outcomes via plain X-ray of pelvis showing both hips through anteroposterior, inlet and outlet views. Evaluation of five criteria on X-ray films postoperatively: residual posterior displacement, vertical displacement, pubic symphyseal translation, sagittal rotation and gapping of the sacroiliac joint. According to the grading of Matta & Tornetta principles, results will be as follows; excellent (< 4 mm), good (4 - 10 mm), fair (10- 20 mm), and poor (> 20 mm).
Clinical outcome score | 12 months
  Clinical outcome assessment at final follow up using Majeed pelvic score. Five factors are assessed and scored: pain, standing, sitting, sexual intercourse and work performance. The total score is then given a clinical grade as excellent, good, fair or poor.

SECONDARY OUTCOMES:
Operative time in minutes. | 3 hours
  Operative time will be recorded in each group
Implant failure rate | 12 months
  Implant failure if any, will be recorded during follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided